CLINICAL TRIAL: NCT00424554
Title: A Phase II Trial to Evaluate the Effect of Low Dose Temozolomide (TMZ) for 2 Weeks on Brain Tumor O-6-methylguanine-DNA Methyltransferase (MGMT) Activity in Patients With Gliomas.
Brief Title: Low-dose Temozolomide for 2 Weeks on Brain Tumor Enzyme in Patients With Gliomas (P04602 AM1) (Completed)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04602
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Results first posted 2011-06-29 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Temozolomide treatment (Experimental)
  Interventions: Drug: temozolomide
- No treatment (No Intervention)

INTERVENTIONS:
Drug: temozolomide — Temozolomide 75 mg/m^2 daily for 14 days prior to surgery.
  As standard of care, it could also be given at the same dose for up to 28 days after surgery, per investigator discretion.
  Other Names: SCH 052365
  Arms: Temozolomide treatment

SUMMARY:
The main purpose of this study is to assess the effect of a two-week pre-surgery treatment with low-dose temozolomide (TMZ) on brain tumor methylguanine-DNA (deoxyribonucleic acid) methyltransferase (MGMT) activity in patients with gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a brain tumor with high probability of being a glioma as detected by Magnetic Resonance Imaging (MRI). These would include newly diagnosed tumors or potentially recurrent gliomas.
* No prior treatment for the tumor including chemotherapy or radiotherapy.
* Amenable to surgery for biopsy or resection of the brain tumor. Surgically confirmed diagnosis of glioma (glioblastoma multiforme [GBM], anaplastic astrocytoma [AA], anaplastic oligodendroglioma [AO], anaplastic oligoastrocytoma [AOA], astrocytoma [A] or oligodendroglioma [O]) will be

required for patients to be maintained in the study. Those not fulfilling this requirement will be discontinued and will be replaced.

* Use of medically approved contraception in fertile males and females.
* Women with childbearing potential must have a negative urine or serum

pregnancy test (urinary excretion or serum level of beta-Human Chorionic

Gonadotropin [bHCG]) within 72 hours of randomization.

* Karnofsky Performance Status score >= 70%.
* Signed informed consent form

Exclusion Criteria:

* Prior chemotherapy.
* Prior radiotherapy at the tumor site.
* History of non-compliance to other therapies.
* Inadequate haematological, renal and hepatic function according to all of the following laboratory values (to be performed within 14 days, inclusive, prior to study inclusion):

  * Absolute neutrophil count ≤1.5 x 10^9/L;
  * Platelets ≤100 x 10^9/L;
  * Haemoglobin <90 g/L;
  * Serum creatinine ≥1.5 times upper limit of laboratory normal;
  * Total serum bilirubin ≥1.5 times upper limit of laboratory normal (ULN);
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.0 ULN;
  * Alkaline phosphatase of > 2.5 ULN.
* Known Human Immunodeficiency Virus [HIV] infection.
* Known chronic hepatitis B or hepatitis C infection.
* Any other serious medical condition according to the medical judgment of the physician prior to inclusion in the study.
* Any medical condition, which could interfere with oral medication intake (e.g., frequent vomiting, partial bowel obstruction).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-09-26 (Actual); Primary Completion 2010-01-11 (Actual); Study Completion 2011-02-16 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Temozolomide (TMZ): Temozolomide 75 mg/m^2 daily for 14 days prior to surgery.
  As standard of care, it could also have been given at the same dose for up to 28 days after surgery, per investigator discretion.
- No Intervention: No pre-surgery treatment with temozolomide
Period: Overall Study
Arm/Group | Temozolomide (TMZ) | No Intervention
Started | 34 | 6
Completed | 34 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Temozolomide (TMZ) | No Intervention | Total
Number analyzed (Participants) | 34 | 6 | 40
Age, Customized [Number; unit: Participants] — Age range: 18-75 years
  Participants | 34 | 6 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 4 | 21
  Male | 17 | 2 | 19
Region of Enrollment [Number; unit: participants]
  Canada | 34 | 6 | 40

OUTCOME MEASURES:

1. Primary Outcome: MethylGuanine-DNA MethylTransferase [MGMT] Activity Measured From the Tumor Tissue During Surgery
Description: An experimental assay was developed to measure MGMT levels.
Time Frame: 14 days
Population: All participants for which a MGMT activity assay could be
  performed
Measure: Mean (Standard Deviation); unit: fmol/mg of proteins
Arm/Group | Temozolomide (TMZ) | No Intervention
Number analyzed (Participants) | 33 | 5
fmol/mg of proteins | 333.7 (288.5) | 105.1 (155)
Statistical Analysis 1: Comparison: Temozolomide (TMZ) vs No Intervention; Test type: Superiority or Other; p = 0.09, t-test, 2 sided

2. Secondary Outcome: Safety: Number of Participants Who Experienced Grade 3 or 4 Toxicities
Description: Grade 3 was defined as severe per Common Terminology Criteria for Adverse Events (CTCAE).
  Grade 4 was defined as life-threatening per CTCAE.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Temozolomide (TMZ) | No Intervention
Number analyzed (Participants) | 34 | 6
participants
  Grade 3 | 4 | 0
  Grade 4 | 0 | 0

3. Secondary Outcome: Tolerability: Number of Participants Discontinuing Treatment Due to Adverse Events (AE)
Description: An AE was defined as any event which was adverse, including what were commonly described as adverse or undesirable experiences, adverse events, adverse reactions, side effects, or death due to any cause associated with, or observed in conjunction with the use of a drug, biological product, or device in humans, whether or not considered related to the use of that product. Additionally, any event which was associated with, or observed in conjunction with product overdose whether accidental or intentional, or product abuse and/or withdrawal was also considered an AE.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Temozolomide (TMZ) | No Intervention
Number analyzed (Participants) | 34 | 6
participants | 0 | 0

4. Secondary Outcome: Concentrations of Temozolomide in the Serum, Cerebrospinal Fluid, and Brain Tumor
Description: No data available: at the time of tumor collection, the temozolomide levels were below the detection limits of the assay.
Time Frame: 14 days
Arm/Group | Temozolomide (TMZ) | No Intervention
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: MGMT Activity in the Brain Tumor Tissues by Temozolomide Levels
Description: as for outcome 4
Time Frame: 14 days
Arm/Group | Temozolomide (TMZ) | No Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Temozolomide: Temozolomide 75 mg/m^2 daily for 14 days prior to surgery.
  As standard of care, it could also have been given at the same dose for up to 28 days after surgery, per investigator discretion.
Arm/Group | Temozolomide | No Intervention
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/6
Other Adverse Events (participants affected / at risk) | 13/34 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=34) | No Intervention (N=6)
LYMPHOPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1)
POSTOPERATIVE FEVER (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
COMPLEX PARTIAL SEIZURES (Nervous system disorders) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 0 (0) | 1 (2)
HEMIPARESIS (Nervous system disorders) | 2 (2) | 1 (1)
SPEECH DISORDER (Nervous system disorders) | 1 (1) | 1 (1)
VISUAL FIELD DEFECT (Nervous system disorders) | 4 (4) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The assay developed to measure MGMT activity had high variability.

The TMZ assay was unable to detect the low levels of the drug due to the relatively low dose and short half life of TMZ.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator (PI) agrees not to publish or publicly present any interim results of the Study without prior written consent of the sponsor. The PI further agrees to provide 45 days written notice to the sponsor prior to submission for publication or presentation to permit the sponsor to review, without limitation, including editorial rights. If the parties disagree, the PI agrees to meet with the sponsor to discuss and resolve any such issues or disagreement.